CLINICAL TRIAL: NCT02983097
Title: Open-label, Multicenter Phase I/II Study: Salvage Therapy of Progressive and Relapsed Aggressive Non-Hodgkin-Lymphoma by Combination of Lenalidomide (Revlimid®) With Rituximab, Dexamethason, High-dose ARA-C and Cisplatinum (R²-DHAP)
Brief Title: Therapy of Non-Hodgkin-Lymphoma by Combination of Lenalidomide + Rituximab, Dexa, High-dose ARA-C and CisP
Acronym: R²-DHAP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase II: no scientific interests are given anymore
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: Celgene (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2008 R6; 2009-010824-25 (EudraCT Number)
Record Dates: First submitted 2013-11-14; First posted 2016-12-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2016-12

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL); Follicular Lymphoma Grade III (FL III°); Mantle Cell Lymphoma (MCL), Blastoid Variant; Burkitt Lymphoma (BL); Aggressive Marginal Zone Lymphoma (MZL)
Keywords: lymphoma; relapse; recurrence; progress; progressive; b-cell lymphoma; chemotherapy; immunotherapy; IMiD; Salvage chemotherapy; peripheral stem cell mobilization; lenalidomide; Rituximab; CD20; Cytarabine; Ara-C; platinum-based chemotherapy; Cisplatin; Carboplatin; Cisplatinum; Carboplatinum; Dexamethasone
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma; Recurrence; Lymphoma, B-Cell | interventions — Rituximab; Cisplatin; Carboplatin; Dexamethasone; Cytarabine; Lenalidomide; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R²-DHAP (Experimental): Combination treatment with immunochemotherapy (R-DHAP) and lenalidomide
  Dosage:
  Rituximab 375 mg/m² day 1, i.v. Cisplatin 100 mg/m² or Carboplatin AUC5 day 2, i.v. Cytarabine 2000 mg/m², administered twice, on day 3, i.v. Dexamethasone 40 mg, days 2-5, p.o. Lenalidomide 5-20 mg, day 1-7 / day-6-+7, p.o. PEG-Filgrastim 6 mg, day 6, s.c.
  peripheral stem cell collection after cycle 1 or 2
  Interventions: Drug: Rituximab; Drug: Cisplatin; Drug: Carboplatin; Drug: Dexamethasone; Drug: Cytarabine; Drug: Lenalidomide; Drug: PegFilgrastim; Procedure: peripheral stem cell collection

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m²
  Other Names: MabThera
Drug: Cisplatin — Cisplatinum 100 mg / m²
  Other Names: Cisplatinum
Drug: Carboplatin — Carboplatinum AUC5
  Other Names: Carboplatinum
Drug: Dexamethasone — Dexamethasone 40 mg
Drug: Cytarabine — Cytarabine 2000 mg/m², administered twice
  Other Names: Cytarabin; Ara-C
Drug: Lenalidomide — 5-20 mg administered either d1-d7, or d-6-d7
  Other Names: Revlimid
Drug: PegFilgrastim — PegFilgrastim 6 mg
  Other Names: Neulasta
Procedure: peripheral stem cell collection — collection of peripheral stem cells for autologous stem cell transplantation
  Other Names: peripheral stem cell apheresis; hematopoetic stem cell apheresis; peripheral hematopoetic stem cell apheresis

SUMMARY:
The goal of this study is to evaluate efficacy and safety of the combination of lenalidomide, an immunomodulatory drug (IMiD) with a standard immunochemotherapy treatment, called R-DHAP. R-DHAP consists of a monoclonal antibody called Rituximab and chemotherapy consisting of Dexamethasone, high dose Cytarabine, often called Ara-C, and platinum based chemotherapy, either cisplatinum, or, if treatment with cisplatinum is contraindicated, carboplatinum.

DETAILED DESCRIPTION:
This is a phase 1/2 study to evaluate the efficacy and safety of lenalidomide added to a standard chemotherapy regime of R-DHAP (Rituximab, Dexamethasone, high-dose Cytarabine, Cis/Carboplatinum) in the treatment of relapsed or refractory high-grade B-cell non-hodgkin-lymphoma (NHL).

The study hypothesis is that the combination of lenalidomide with standard immunochemotherapy will lead to an overall response rate of at least 60%. In this study, 3 rounds of immunochemotherapy in combination with lenalidomide will be administered. After the first or second round of therapy, peripheral hematopoetic stem cells will be harvested. Consolidation treatment with autologous or allogenic peripheral blood stem cell transplantation is recommended in all patients suitable, but is not part of the study.

In phase 1, up to six cohorts of at least 6 patients each will be treated with the study therapy, with lenalidomide in increasing dosages, to determine the maximum tolerated dose (MTD).

In phase 2, 50 patients will be treated with the MTD. Efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-70

Risk groups: All risk groups

histology: diagnosis or a recurrent or primary progressive aggressive b-cell non-hodgkin lymphoma, in particular

* follicular lymphoma grade III
* diffuse large b-cell lymphoma
* burkitt lymphoma
* mantle cell lymphoma, blastoid variant
* aggressive marginal zone lymphoma

Performance status: ECOG 0-2

Criteria for women of childbearing potential:

Women of childbearing potential have to:

* understand the teratogenic risk associated with the study therapy, especially lenalidomide
* understand the need of reliable, uninterrupted birth control from 4 weeks prior to the start of the study drug, during the duration of the study treatment, and 4 weeks after completion of study treatment, and be able to reliably use birth control, except if the patient commits to absolute sexual abstinence, confirmed on a monthly basis

The following are effective methods of contraception:

* implant
* levonorgestrel-releasing intrauterine system (IUS)
* medroxyprogesterone acetate depot
* tubal sterilisation
* sexual intercourse with a vasectomised male partner only, vasectomy must be confirmed by two negative semen analyses
* ovulation-inhibitory progesterone-only pills If not established on effective contraception, the female subject must be referred to an appropriately trained health care professional for contraceptive advice in order that contraception can be initiated.
* Understand that even if she has amenorrhea, she must follow all the advice on effective contraception
* Understand the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy.
* Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml on the day of the study visit or in the 3 days prior to the study visit once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence. The test should ensure the subject is not pregnant when she starts treatment.
* Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These pregnancy tests should be performed on the day of the study visit or in the 3 days prior to the study visit. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.

Male patients have to:

* Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
* Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.

All patients have to:

* Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
* Agree not to share study medication with another person and to return all unused study drug to the investigator

Patients must be able to take low molecular weight heparin as prophylactic anticoagulation

Written informed consent is necessary

Exclusion Criteria:

* pregnant or lactating females
* already initiated salvage lymphoma therapy (except prephase as specified in this study)
* serious accompanying disorder or impaired organ function causing significant clinical problems and reduced lyfe expectancy, in particular: heart: angina pectoris CCS>2 cardiac failure NYHA>2 and/or EF<45% lungs: FeV1<60%, diffusion capacity <50% of the reference values kidneys: creatinine>2 times the upper reference limit liver: bilirubin >2 times the upper reference limit
* platelets <80000/mm³, leukocytes <2500/³
* CNS involvement of lymphoma
* known hypersensitivity to the medications to be used
* known HIV-positivity
* suspicion that patient compliance will be poor, especially that rules for effective contraception will not be followed
* simultaneous participation in other treatment studies
* non-conformity to eligibility criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2015-04-28 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 78 - 85 days + 2 years Follow Up
  The percentage of patients which showed either a partial remission (PR), a complete remission with remaining uncertainty (CRu) or a complete remission (CR) after study treatment.
Maximum tolerated dose (MTD) | 78 - 85 days
  The maximum dose of lenalidomide tolerated with acceptable toxicity during phase 1 of this study. The MTD established in phase 1 of this study will be administered to 50 patients in phase 2 of this study.

SECONDARY OUTCOMES:
Rate of complete remission | 78 - 85 days + 2 years Follow Up
  laboratory, BM biopsy, imaging
Rate of primary progression | 78 - 85 days + 2 years Follow Up
  The rate of patients which show progressive disease (PD) during or directly after study therapy
Rate of treatment related deaths | 78 - 85 days + 2 years Follow Up
  check survival
Relapse Rate | 78 - 85 days + 2 years Follow Up
  laboratory, BM biopsy, imaging
Overall Survival | 78 - 85 days + 2 years Follow Up
  check survival
Progression free survival | 78 - 85 days + 2 years Follow Up
  laboratory, BM biopsy, imaging
tumour control | 78 - 85 days + 2 years Follow Up
  laboratory, BM biopsy
feasibility of stem cell mobilization | 78 - 85 days + 2 years Follow Up
  The collection of peripheral stem cells is needed to be able to offer the patient high dose chemotherapy followed by autologous stem cell transplantation after the study treatment has ended.
  Stem cell collection of <2.0 *10e6 CD34+cells/kg will be considered insufficient.
incidence of non-hematological toxicities > grade 2 CTC | 78 - 85 days + 2 years Follow Up
incidence and duration of neutropenia and thrombopenia grade 4 | 78 - 85 days + 2 years Follow Up
  laboratory WBC < 1.0 /nl or Plt < 25 /nl

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Glaß, MD, Principal Investigator — AK St.Georg
Locations (12):
- Germany (12):
  - Diakonie Krankenhaus Bremen, Bremen
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Essen, Essen
  - Klinikum Frankfurt/Oder, Frankfurt (Oder)
  - Universitätsklinikum Göttingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Westpfalz Klinikum, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - LMU Klinikum München-Großhadern, München

REFERENCES:
- See also: Homepage of the "Kompetenznetz Maligne Lymphome" — http://www.lymphome.de/